CLINICAL TRIAL: NCT05675592
Title: Linking Elexacaftor/Tezacaftor/Ivacaftor to Infections in Cystic Fibrosis Lung Disease
Brief Title: Trikafta/Kaftrio and Pseudomonas Aeruginosa
Acronym: Kaf-Pseudo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Ospedale Pediatrico Bambin Gesù (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Cristina Cigana, Research Associate - Principal Investigator, Ospedale San Raffaele
Other Study IDs: 173/INT/2021; FFC#16/2021 (Other Grant/Funding Number: Italian Cystic Fibrosis Research Foundation)
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Cystic Fibrosis
Keywords: Trikafta; Pseudomonas aeruginosa; susceptibility to antibiotics; bacterial phenotype; bacterial transcriptome; bacterial genome; bacterial virulence
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Pseudomonas aeruginosa strains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study o is to define whether, how and to what extent treatment with Trikafta/Kaftrio directly affects Pseudomonas aeruginosa in individuals with cystic fibrosis. The main questions it aims to answer are:

* whether Trikafta/Kaftrio affects the bacterial phenotypes and susceptibility to antibiotics;
* whether Trikafta/Kaftrio impacts the bacterial virulence. Participants will be asked the permission to store and analyze P. aeruginosa isolates collected from respiratory samples for usual care plans before the initiation of treatment with Trikafta/Kaftrio and after 12 and 18 months of treatment. The results of bacterial analysis will be matched with clinical data at the specific time-points.

We expect to define effects of Trikafta/Kaftrio on P. aeruginosa and identify bacterial phenotypes as possible risk factors for its efficacy.

DETAILED DESCRIPTION:
We will recruit 20 individuals affected by cystic fibrosis (≥12 years of age), chronically infected with P. aeruginosa (defined as having at least 50% or more sputum cultures positive for P. aeruginosa in the previous year), homozygous for the F508del mutation (F508del/F508del) or heterozygous for the F508del mutation and with a minimal function mutation in the other allele (F508del/minimal function), candidates for treatment with Trikafta/Kaftrio according to clinical practice. P. aeruginosa strains will be collected from the sputum before the start of therapy (T0) and after 12 (T12m) and 18 (T18m) months of treatment with Trikafta/Kaftrio. Currently, some patients have already started treatment with Trikafta/Kaftrio. The strains at T0 and for some of them also at T12m and T18m have already been recovered from these patients for other studies. Of these strains it is not yet known whether they are clonal at different times (T0, T12m and T18m). Of these patients, we will include in the expected 20 (20 total between prospective and retrospective) only patients for whom strains clonal between T0, T12m and T18m will be identified, asking for their authorization to use the strains and their data through informed consent. If the number of retrospective patients is sufficient to reach the expected number (20 total patients), no other patients will be recruited prospectively.

Patients who will be prescribed Trikafta/Kaftrio therapy according to clinical practice will be recruited at routine visits. The decision to prescribe treatment with Trikafta/Kaftrio, according to current clinical practice, is completely independent of the decision to include the patient in this study. The diagnostic and evaluation procedures and follow-up visits foreseen by the study will coincide with those programmed for each patient according to the standard operating procedures in force at the participating centres.

For retrospective patients, informed consent will be collected during the routine check-up and, once the eligibility criteria have been verified, the data relating to the visit performed before the start of therapy (T0) and, if already available, the data relating to the visit performed at 12 and 18 months from the beginning of the therapy (T12m and T18m), will be collected. P. aeruginosa recovered from the respiratory samples during the three visits will be analysed. In the event that data are not available, data and samples will be collected at the respective routine follow-ups (at 12 and/or 18 months).

For prospective patients, the enrollment visit will be performed during the routine visit performed before the start of therapy (T0) which will be followed by visits scheduled for clinical practice at 12 and 18 months from the start of therapy (T12m and T18m).

At T0, T12m and T18m the sputum samples, collected from the patient's airways, will be treated according to standard procedures for the evaluation of the bacterial species present. P. aeruginosa strains will be subjected to minimal inhibitory concentration tests to assay their susceptibility to a panel of standard antibiotics, and analyzed by Multi-locus Sequence Typing to detect their clonality.

The strains of each patient that will be clonal between T0, T12m and T18m, immediately stored at -80°C, will then be shipped to Ospedale San Raffaele , where they will be analyzed for the purposes of the project using methods validated in the literature. We will analyze i) the phenotypes (in particular motility by pilus, motility by flagellum, secretion of proteases and pyocyanin, and mucoidity) of P. aeruginosa strains using microbiological methods validated in the literature, ii) the expression profiles of the strains by RNA sequencing, iii) the presence of gene variants by whole genome sequencing of the strains, iv) and their virulence by measuring their impact on the expression of the cystic fibrosis transmembrane conductance regulator protein in cystic fibrosis bronchial epithelial cell lines.

The final aim will be to i) evaluate the differences in the phenotypes of the P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m post treatment with Kaftrio; ii) to evaluate differences in the susceptibility to antibiotics of the P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m; iii) evaluate differences in the expression profiles of the P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m and correlate them to the difference in respiratory function measured as FEV1 (%); iv) evaluate the presence of gene variants between the strains isolated at T0 and those isolated at T12m and T18m and correlate them to the difference in respiratory function measured as FEV1 (%); v) to determine whether changes in bacterial phenotypes induced by Kaftrio treatment may be associated with lower anti-CFTR activity of P. aeruginosa.

ELIGIBILITY:
Inclusion Criteria:

* Definite diagnosis of CF and regular follow up, in accordance with the standard operating procedures in force at the Centres
* Homozygous for the F508del mutation (F508del/F508del) in the CFTR gene or heterozygous for the F508del mutation and with a minimal function mutation in the other allele (F508del/minimum function mutation)
* Chronically infected with P. aeruginosa (defined as having at least 50% or more sputum cultures positive for P. aeruginosa in the previous year)
* Candidates starting treatment with Kaftrio or being treated with Kaftrio (retrospective phase)
* Both sexes aged >12 years
* Obtaining informed consent from patients and/or from patients' parents (according to the modalities foreseen by the protocol)

Exclusion Criteria:

* Patients unable to understand the instructions and information provided and to be able to adequately accept the modalities of the study.
* Patients unable to expectorate.
* Patients with negative sputum for P. aeruginosa at T0, which in the case of prospective patients corresponds to the time of enrollment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 patients with CF (from IRCCS Ca' Granda Foundation, Ospedale Maggiore Policlinico, Milan; IRCCS Pediatrico Bambino Gesù, Rome) will be enrolled. Currently, some patients already started treatment with Kaftrio and P. aeruginosa strains have been recovered for other studies. Of these patients, we will include only those for whom clonal strains at T0, T12m and T18m will be identified. If the number of retrospective patients is sufficient, no other patients will be recruited prospectively.
  Once enrolled, patients may drop out of the study if:
  1. they are unable to expectorate at T12m and T18m;
  2. the sputum is negative for P. aeruginosa at T12m or T18m;
  3. none of the P. aeruginosa strains isolated at T12m and T18m is clonal to at least one strain isolated at T0.
  If the dropout is higher than expected, recruitment will continue until the necessary number of samples to be analyzed is obtained.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-11-16 (Estimated); Study Completion 2025-05-16 (Estimated)

PRIMARY OUTCOMES:
bacterial phenotypes | 0-18 months
  motility by pilus, motility by flagellum, secretion of proteases, secretion of pyocyanin of P. aeruginosa strains isolated at T0 and clonal ones isolated at T12m and T18m post treatment with Trikafta/Kaftrio
respiratory function | 0-18 months
  respiratory function, evaluated as FEV1 (%), measured at time at T0, T12m and T18m post Trikafta/Kaftrio treatment

SECONDARY OUTCOMES:
susceptibility to antibiotics | 0-18 months
  susceptibility of P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m to standard antibiotics evaluated by minimal inhibitory concentration assays
mucoidy | 0-18 months
  mucoidy of the P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m determined by visual assessment of the growth in the plate
expression profile | 0-18 months
  expression profiles of the P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m evaluated by RNA sequencing
genetic variants | 0-18 months
  presence of gene variants, identified by whole genome sequencing, between the strains isolated at T0 and those isolated at T12m and T18m
impact on CFTR | 0-18 months
  Membrane expression of CFTR protein, measured by western blot, in FC and non-FC immortalized bronchial epithelial cell lines stimulated with growth media of P. aeruginosa strains isolated at T0 and those isolated at T12m and T18m

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - UOC Pediatria Fibrosi Cistica, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico, Milan
  - UOC Fibrosi Cistica, IRCCS Ospedale Pediatrico Bambino Gesù, Rome

IPD SHARING:
Plan to Share IPD: Undecided
We are going to discuss this issue

REFERENCES:
- See also: project behind this study — https://www.fibrosicisticaricerca.it/progetto/ffc-16-2021-valutazione-delle-proprieta-antibatteriche-del-kaftrio/